CLINICAL TRIAL: NCT05253365
Title: French Memory Support System: A Pilot Study / Un Systeme de Support de Memoire en Francais: Une Etude de Faisabilite
Brief Title: French Memory Support System: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: M16-21-035
Record Dates: First submitted 2022-01-04; First posted 2022-02-23 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Mild Cognitive Impairment
Keywords: cognition; french
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Memory Support System participants (Experimental)
  Interventions: Behavioral: Memory Support System

INTERVENTIONS:
Behavioral: Memory Support System — The MSS is a two-page-per-day, pocket-sized calendar/note-taking system with three sections: (a) events; (b) to do's; and (c) journaling for logging important things to be remembered (e.g., news about family/friends). MSS training consists of ten 1-hour sessions delivered over two or six weeks, starting 7-10 days after baseline assessment.

SUMMARY:
The purpose of this study is to develop a linguistically and culturally appropriate adaptation of the Memory Support System (MSS), an evidence-based intervention to train persons with mild cognitive impairment (MCI) to complete personal goals and instrumental activities of daily living independently. The study will involve development of the associated manual, training and patient forms, and outcome measures, and pilot testing of the intervention in a group of French-speaking individuals with MCI and their care partners

DETAILED DESCRIPTION:
At enrollment, participants with MCI and their care partners will complete French measures evaluating cognitive and functional status. Participants and partners will also complete French measures of treatment adherence, instrumental activities of daily living, self-efficacy for memory, quality of life, mood, anxiety, and caregiver burden at baseline, treatment end, and 8-week follow-up. Participants will complete the MSS training consisting of ten 1-hour sessions delivered over two or six weeks, starting 7-10 days after initial assessment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of single or multi-domain MCI
* Clinical Dementia Rating global (CDR) score of ≤ 0.5
* Dementia Rating Scale-Second edition score of ≥ 115
* available contact with a care partner ≥ 2 times weekly
* absence or stable intake of nootropic(s) for ≥ 3 months

Exclusion Criteria:

* visual/hearing impairment and/or history of reading or written inability/disability sufficient to interfere with MSS training
* concurrent participation in another related clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Adherence to French Memory Support System Intervention | One week after starting the treatment (MSS intervention), treatment end, and at 8 week follow-up after treatment end.
  Change from adherence scores from one week after starting treatment (MSS intervention) at treatment end and at 8 weeks after the treatment end. Using an adherence scale from 0 to 10, with 10 being highest and a cut-off score of ≥ 7 points suggesting adherence with the MSS.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale | Baseline, treatment end and at 8 week follow-up.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Depression screening scale using Likert scale. Total score of 0-60 points, with higher scores signifying a worse outcome (higher levels of depression).
Everyday Cognition questionnaire. | Baseline and at 8 week follow-up.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Self report measure of performance based instrumental activities of daily living. Total score of 23-92, with higher scores indicating a worse outcome.
Functional Assessment Questionnaire | Baseline and at 8 week follow-up.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Informant based report of performance of instrumental activities of daily living. Total score of 0-30, with higher scores indicating a worse outcome (higher level of dependence).
Quality of Life in Alzheimer Disease | Baseline and at 8 week follow-up.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Self report quality of life scale. Total score of 13-52, with higher scores indicating a better outcome (better quality of life).
State-Trait Anxiety Inventory by the Resources for Enhancing Alzheimer's Caregiver Health project | Baseline and at 8 week follow-up.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Self report anxiety scale. Total score of 10-40 with higher scores indicating a worse outcome (higher level of anxiety).
Chronic Disease Self-efficacy Scale | Baseline and at 8 week follow-up.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Selected questions related to memory and cognition from self report scale. Total score of 9-90 with higher scores indicating a better outcomes (higher feeling of self-efficacy).
Caregiver Burden Inventory Short-Form | Baseline and at 8 week follow-up.
  Change from baseline scale scores at treatment end and at 8 weeks after treatment end. Informant based scale of level of caregiver burden. Total score of 0-48 with higher scores indicating a worse outcome (higher level of burden).

CONTACTS AND LOCATIONS:
Overall Officials: Neil W Thomas, MD, Principal Investigator — Bruyère Health Research Institute.; Octavio Santos, PhD, Principal Investigator — Ottawa Hospital Research Institute, Bruyere Research Institute
Locations (1):
- Bruyere Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No